CLINICAL TRIAL: NCT04259580
Title: Calgary Registry for Advanced and Therapeutic Endoscopy
Acronym: CReATE
Status: Recruiting | Type: Observational
Sponsor: University of Calgary (Other)
Responsible Party: Sponsor
Other Study IDs: REB18-0410
Record Dates: First submitted 2020-02-04; First posted 2020-02-06 (Actual); Last update posted 2024-12-20 (Actual); Status verified 2024-12

CONDITIONS: Biliary Disease; Pancreatic Diseases
MeSH Terms: conditions — Gallbladder Diseases; Pancreatic Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Procedure: Endoscopic retrograde pancreatography (ERCP) — Endoscopic procedure to access biliary and/or pancreatic structures

SUMMARY:
The aim of the Calgary Registry for Advanced and Therapeutic Endoscopy (CReATE) is to be a high-fidelity prospective multi-centre registry. The study population consists of consecutive adult ERCP patients from September 2018 to August 2022. Informed consent is acquired for each patient. All relevant pre-procedural, procedural, peri-procedural and post-procedural data are captured in real time by a full-time third-party research assistant directly observing procedures. Outcomes are ascertained by comprehensive medical record review and patient phone interview 30 days after the index procedure. This registry also serves as a secure data collection platform for several currently recruiting prospective studies and randomized trials.

ELIGIBILITY:
Inclusion Criteria:

* any standard indication for ERCP, in the absence of standard contraindications;
* age 18 years or over;
* ability and willingness to give informed consent to be included in the registry and/or to involvement in one (or more) prospective sub-studies, or accompaniment by a surrogate who is willing and able to provide consent.

Exclusion Criteria:

-none other than inverses of above.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult patients undergoing ERCP.
Sampling Method: Non-Probability Sample
Enrollment: 6000 (Estimated)
Dates: Start 2018-09-01 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Rate of unplanned healthcare utilization | 30 days
  Composite outcome of post-ERCP pancreatitis, bleeding, cholangitis or sepsis, or any other adverse event deemed related to the index procedure, or emergency department presentation or inpatient admission within 30 days deemed related to the index procedure.

SECONDARY OUTCOMES:
Rate of post-ERCP pancreatitis | 30 days
  Typical abdominal pain with amylase/lipase 3 times normal or higher
Rate of post-ERCP bleeding | 30 days
  Hematemesis and/or melena or hemoglobin drop 2 g or greater
Rate of post-ERCP cholangitis or sepsis | 30 days
  Fever > 38C for 24 hours or more with cholestasis, or positive blood cultures
Technical success rates | Immediate

CONTACTS AND LOCATIONS:
Locations (1):
- University of Calgary, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: Yes
Future studies will utilize patient-specific data, which will be in a de-identified encrypted secure format whenever shared.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: For 5 years after data collection is complete.

REFERENCES:
- [Derived] Mohamed R, Lethebe BC, Gonzalez-Moreno E, Kayal A, Bass S, Cole M, Turbide C, Chau M, Koury HF, Brenner DR, Hilsden RJ, Elmunzer BJ, Keswani RN, Wani S, Heitman SJ, Forbes N. Morphology of the major papilla predicts ERCP procedural outcomes and adverse events. Surg Endosc. 2021 Dec;35(12):6455-6465. doi: 10.1007/s00464-020-08136-9. Epub 2020 Nov 4. PMID 33146812